CLINICAL TRIAL: NCT03384446
Title: The Role of Dental Hygiene Procedures in Disruption of Healthy Homeostasis in Tissues Surrounding Dental Implants - Phase I
Brief Title: Dental Hygiene and Peri-Implant Tissues Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Osteogenics Biomedical (Industry)
Responsible Party: Principal Investigator, Giorgios Kotsakis, Assistant Professor, School of Dentistry:Dept. of Periodontics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002852
Record Dates: First submitted 2017-12-19; First posted 2017-12-27 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which intervention was administered. Outcome assessor will be different than care provider and will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth-borne treatment (Active Comparator): A cleaning aid that resembles tooth cleaning instruments and is empirically used for implant surface cleaning.
  Interventions: Other: Tooth-borne treatment
- Implant-specific treatment (Experimental): A cleaning aid that has been specifically designed for implant surface cleaning.
  Interventions: Other: Implant-specific treatment

INTERVENTIONS:
Other: Tooth-borne treatment — Titanium curettes
  Arms: Tooth-borne treatment
Other: Implant-specific treatment — Implant brush
  Arms: Implant-specific treatment

SUMMARY:
Dental implants have revolutionized the field of dentistry, providing improvements in function and esthetics. They are not, however, without risks. Bone loss around implants (i.e. periimplantitis) is an emerging public health concern. Untreated, peri-implantitis leads to implant loss and jawbone defects. Nonetheless, existing therapies have failed to show long-term efficacy. The pathogenesis of peri-implantitis is believed to be of bacterial etiology similar to periodontal disease. Therefore, existing treatments duplicate strategies for the treatment of natural teeth. However, the titanium (Ti) surface of implants is quite dissimilar to teeth. Recent work from our lab has demonstrated that peri-implantitis is associated with increased release of Ti particles around implants. These findings suggest that treatments targeting periimplantitis must be designed around Ti material properties. A gap in knowledge exists regarding the potential triggers of increased Ti dissolution from the implant surface and the mechanisms by which Ti dissolution products amplify peri-implant inflammation. The aim of this study is to determine if the use of tooth-driven treatment approaches increase Ti in the submucosal plaque.

ELIGIBILITY:
Inclusion Criteria:

* Is the subject ≥ 25 years of age?
* Does the subject have an implant with a probing depth ≥ 5mm, bleeding on probing, and radiographic bone loss of > 2mm?
* Is the subject committed to the study and the required follow-up visits?

Exclusion Criteria:

* Is the subject immune compromised?
* Is the subject diabetic?
* Does the subject take steroid medication?
* Does the subject regularly use non-steroidal anti-inflammatories?
* Is the subject pregnant or intending to become pregnant during the duration of the study?
* Has the subject had previous implantoplasty?
* Did the subject take any antibiotics in the last 3 months?

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Titanium elution | 8 weeks
  The primary outcome of the clinical trial will be titanium dissolution in periimplant plaque at 8 weeks following treatment quantified using inductively coupled mass spectrometry (ICMS)

SECONDARY OUTCOMES:
Probing depth reduction | 5 months, 12 months
  Probing depth reduction following surgical peri-implant treatment
BOP reduction | 5 months, 12 months
  Changes in % bleeding on probing following surgical peri-implant treatment
Bone level changes | 5 months, 12 months
  Changes in peri-implant bone level as assessed via standardized radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Kotsakis, DDS, MS, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - UTHealth San Antonio, San Antonio, Texas
  - University of Washington, Department of Periodontics, Seattle, Washington

REFERENCES:
- [Result] Daubert D, Lee E, Botto A, Eftekhar M, Palaiologou A, Kotsakis GA. Assessment of titanium release following non-surgical peri-implantitis treatment: A randomized clinical trial. J Periodontol. 2023 Sep;94(9):1122-1132. doi: 10.1002/JPER.22-0716. Epub 2023 May 2. PMID 37070363